CLINICAL TRIAL: NCT06690216
Title: Evaluation of the Value of [18F]AlF-NOTA-PCP2 PET/CT for PD-L1 Detection in Malignant Tumors
Brief Title: Evaluation of [18F]AlF-NOTA-PCP2 PET/CT for PD-L1 Detection in Malignant Tumors
Acronym: PD-L1-PET
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Man Hu (Other)
Responsible Party: Sponsor-Investigator, Man Hu, Chief physician, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ShandongCHI202410074; KY-2024-136 (Other: Shandong Cancer Hospital and Institute Shandong First Medical University and Shandong Academy of Medical Sciences: Shan)
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma (GBM); Head and Neck Squamous Cell Carcinoma; Non-Small Cell Lung Cancer; Esophageal Cancer
Keywords: PET/CT; PD-L1 expression; [18F]AlF-NOTA-PCP2; Glioblastoma; Head and neck squamous cell carcinoma; Non-small cell lung cancer; Esophageal cancer; Immunotherapy guidance; Tumor biomarker imaging
MeSH Terms: conditions — Glioblastoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase I/II, single-center, interventional clinical trial assessing the safety, efficacy, and prognostic value of [18F]AlF-NOTA-PCP2 PET/CT in evaluating PD-L1 expression in patients with malignant tumors. The study involves pre-treatment imaging with [18F]AlF-NOTA-PCP2 PET/CT, followed by correlation with PD-L1 expression in tumor samples and clinical outcomes.
Masking Description: This study is open-label, with no masking of any parties involved in the clinical trial. All participants, care providers, investigators, and outcomes assessors are aware of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F]AlF-NOTA-PCP2 PET/CT Imaging for PD-L1 Expression in Malignant Tumors (Experimental): This arm involves the administration of [18F]AlF-NOTA-PCP2 via intravenous injection followed by whole-body PET/CT imaging one hour later. The objective is to assess the uptake of [18F]AlF-NOTA-PCP2 in malignant tumors and correlate it with PD-L1 expression. This imaging technique is used to evaluate PD-L1 expression in glioblastoma, head and neck squamous cell carcinoma, non-small cell lung cancer, and esophageal cancer patients before treatment, providing a non-invasive, repeatable, and comprehensive approach to guide immunotherapy decisions.
  Interventions: Diagnostic Test: PET/CT （[18F]AlF-NOTA-PCP2）; Diagnostic Test: [18F]AlF-NOTA-PCP2 PET/CT Imaging for PD-L1 Expression in Malignant Tumors

INTERVENTIONS:
Diagnostic Test: PET/CT （[18F]AlF-NOTA-PCP2） — This intervention involves the use of [18F]AlF-NOTA-PCP2, a radiopharmaceutical agent specifically designed for PET/CT imaging. Patients will receive an intravenous injection of [18F]AlF-NOTA-PCP2, followed by whole-body PET/CT scanning one hour later. The primary purpose of this intervention is to assess PD-L1 expression in malignant tumors, including glioblastoma, head and neck squamous cell carcinoma, non-small cell lung cancer, and esophageal cancer, before the initiation of treatment. This imaging technique offers a non-invasive, repeatable, and comprehensive method to monitor PD-L1 status, in contrast to traditional tissue biopsy, which is invasive and limited to a single time point.
Diagnostic Test: [18F]AlF-NOTA-PCP2 PET/CT Imaging for PD-L1 Expression in Malignant Tumors — This intervention involves the use of [18F]AlF-NOTA-PCP2, a radiopharmaceutical agent specifically designed for PET/CT imaging. Patients will receive an intravenous injection of [18F]AlF-NOTA-PCP2, followed by whole-body PET/CT scanning one hour later. The primary purpose of this intervention is to assess PD-L1 expression in malignant tumors, including glioblastoma, head and neck squamous cell carcinoma, non-small cell lung cancer, and esophageal cancer, before the initiation of treatment. This imaging technique offers a non-invasive, repeatable, and comprehensive method to monitor PD-L1 status, in contrast to traditional tissue biopsy, which is invasive and limited to a single time point.

SUMMARY:
This phase I/II clinical trial evaluates the safety, efficacy, and prognostic potential of [18F]AlF-NOTA-PCP2 PET/CT imaging in assessing PD-L1 expression in malignant tumors, including glioblastoma, head and neck squamous cell carcinoma, non-small cell lung cancer, and esophageal cancer. The primary aim is to establish the correlation between [18F]AlF-NOTA-PCP2 uptake and PD-L1 expression in tumor tissues, while secondary objectives include evaluating its role in predicting clinical outcomes such as progression-free survival (PFS) and overall survival (OS). By providing a non-invasive, quantitative, and reproducible method for assessing PD-L1, this study aims to refine patient stratification and improve the precision of immunotherapy decision-making.

DETAILED DESCRIPTION:
This phase I/II clinical trial is designed to explore the utility of [18F]AlF-NOTA-PCP2 PET/CT in evaluating PD-L1 expression and its prognostic implications in patients with malignant tumors (glioblastoma, head and neck squamous cell carcinoma, non-small cell lung cancer, and esophageal cancer). The study involves at least 20 patients (5 per tumor type) who will undergo a pre-treatment PET/CT scan following an intravenous injection of [18F]AlF-NOTA-PCP2. The primary endpoints include the safety of the imaging protocol and the correlation between [18F]AlF-NOTA-PCP2 uptake (SUV values) and PD-L1 expression determined through immunohistochemistry (IHC). Secondary endpoints explore the dynamic changes in SUV values in patients undergoing multiple scans and their relationship with clinical outcomes.

Scientific and Technical Rationale:

[18F]AlF-NOTA-PCP2 is a novel radiotracer with high specificity for PD-L1, enabling non-invasive imaging of its expression in vivo. This imaging approach complements traditional immunohistochemical methods by offering whole-body assessment, eliminating the need for repeated biopsies, and providing insights into the tumor microenvironment. This study seeks to validate its application in clinical oncology, bridging molecular imaging with biomarker-guided therapeutic strategies.

Study Methods:

Patients will receive a single intravenous dose of [18F]AlF-NOTA-PCP2 (adjusted for body weight), followed by a whole-body PET/CT scan after one hour. Images will be analyzed independently by two experienced nuclear medicine specialists. Tumor biopsies will be collected to measure PD-L1 expression via IHC, and blood samples will be assessed for circulating and exosomal PD-L1 biomarkers. For patients undergoing multiple scans, changes in radiotracer uptake will be tracked to monitor treatment response.

Data Analysis:

SUV values will be correlated with PD-L1 expression levels, clinical factors (e.g., tumor stage, histology), and patient outcomes (PFS, OS). Statistical analyses, performed using SPSS 29.0, will include primary correlations and secondary evaluations of imaging-based dynamic changes and their relationship with therapeutic efficacy.

Significance:

This trial will provide critical data on the feasibility of [18F]AlF-NOTA-PCP2 PET/CT imaging in clinical oncology. Its potential to stratify patients based on PD-L1 expression and predict therapy response could transform personalized cancer care, optimizing immunotherapy outcomes and minimizing unnecessary treatments.

Timeline:

Patient enrollment is expected to last 12 months, with an additional 3 months of follow-up for data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained.
* Age ≥ 18 years, any gender.
* Pathologically confirmed malignant tumors, including:
* Glioblastoma
* Head and neck squamous cell carcinoma
* Non-small cell lung cancer
* Esophageal cancer
* Detectable PD-L1 expression in tumor tissue (based on immunohistochemistry or biopsy).
* Measurable disease with at least one residual tumor lesion.
* ECOG performance status of 0-1.
* No contraindications to [18F]AlF-NOTA-PCP2 PET/CT imaging.
* Willing and able to comply with study procedures and follow-up visits.

Exclusion Criteria:

* Participation in another interventional clinical trial.
* Failure to recover from toxic effects or complications of prior interventions (≤ grade 1 or baseline levels, excluding fatigue or hair loss).
* Pregnant or breastfeeding women.
* Severe or uncontrolled systemic diseases, including:
* Major, symptomatic arrhythmias or significant ECG abnormalities (e.g., complete left bundle branch block, second-degree or higher heart block, or ventricular arrhythmias).
* Unstable angina or congestive heart failure (NYHA class ≥ 2).
* Any arterial thrombotic or embolic events within 6 months before enrollment (e.g., myocardial infarction, cerebrovascular accident, transient ischemic attack).
* Active or uncontrolled infections requiring systemic treatment.
* Severe psychiatric disorders affecting study participation.
* Any medical history, laboratory abnormality, or condition that may:
* Interfere with study results.
* Affect patient participation.
* Pose an unacceptable risk as determined by the investigator.
* Women of childbearing potential without a negative pregnancy test prior to study entry.
* Known allergy or hypersensitivity to [18F]AlF-NOTA-PCP2 or any component of the radiopharmaceutical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of [18F]AlF-NOTA-PCP2 PET/CT imaging for PD-L1 expression in malignant tumors | Pre-treatment imaging, within 1-7 days before treatment initiation.
  This outcome measure will assess the safety and efficacy of [18F]AlF-NOTA-PCP2 PET/CT in detecting PD-L1 expression in malignant tumors (glioblastoma, head and neck squamous cell carcinoma, non-small cell lung cancer, and esophageal cancer). This will include evaluating the correlation between [18F]AlF-NOTA-PCP2 uptake and PD-L1 expression as determined by immunohistochemistry (IHC).

SECONDARY OUTCOMES:
[18F]AlF-NOTA-PCP2 PET/CT imaging as a prognostic biomarker in malignant tumors | Up to 1 year of follow-up for clinical outcomes (PFS, OS).
  This outcome will evaluate the prognostic value of [18F]AlF-NOTA-PCP2 PET/CT imaging in predicting clinical outcomes, including progression-free survival (PFS) and overall survival (OS), based on tumor PD-L1 expression.

OTHER OUTCOMES:
Correlation of circulating PD-L1 and exosomal PD-L1 with [18F]AlF-NOTA-PCP2 PET/CT imaging | Pre-treatment, and at follow-up visits (up to 1 year).
  This exploratory outcome measure will investigate the correlation between circulating PD-L1 levels, exosomal PD-L1, and [18F]AlF-NOTA-PCP2 PET/CT imaging for assessing PD-L1 expression in tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Man Hu, Dr., Study Chair — Shandong Cancer Hospital and Institute Shandong First Medical University and Shandong Academy of Medical Sciences: Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data (IPD) from this clinical trial, including the following types of data:
  Data to be Shared:
  Demographic Data: Age, sex, and other basic demographic information. Clinical Data: Diagnosis, treatment regimens, disease stage, and clinical outcomes.
  Imaging Data: PET/CT scan images and associated quantitative data (e.g., SUV values) related to [18F]AlF-NOTA-PCP2 uptake.
  Biomarker Data: Results from PD-L1 expression assays, including tissue sample data and blood biomarkers.
  Adverse Event Data: Adverse event reports, including the type, severity, and outcome as graded by the NCI CTCAE.
  How the Data Will Be Shared:
  The IPD will be shared via a secure, password-protected database or a data-sharing platform. Access will be granted to qualified researchers upon submission of a data request proposal.
  The sharing process will include a data use agreement (DUA) that outlines the terms of use, data protection protocols, and the research purposes for which
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: The IPD and supporting information will be available starting after the completion of the primary analysis and publication of study results, which is expected to be by October 2025.
  End Date: The IPD and supporting information will be available for a period of 5 years following study completion, until October 2030.
Access Criteria: Who will have access: Access to the individual participant data (IPD) and supporting information will be available to qualified researchers, healthcare professionals, and institutions involved in academic research or related scientific studies. This may include those interested in replicating the study results, conducting further analyses, or exploring the data for new scientific questions.
  What will be accessible: Researchers will have access to:
  The full individual participant data (IPD), including anonymized data related to clinical outcomes, imaging results (e.g., PET/CT scans), and laboratory tests.
  Supporting documents, such as the study protocol, statistical analysis plan (SAP), informed consent form (ICF), and the clinical study report (CSR), which provide details on the methodology, analysis approach, and results.
  How to access: Researchers can request access to the IPD and supporting information through the official study contact, Dr. Man Hu (contact: mhu@sdfmu.edu.cn). Upo

REFERENCES:
- [Background] Wang Y, Zhang Y, Chen Y, Wang S, Liu W, Liu Z, Hu M. [18F]AlF-NOTA-PCP2: a novel PET/CT tracer for enhanced PD-L1 heterogeneity imaging and comparative analysis with [18F]AlF-NOTA-WL12 in glioblastoma xenografts. Eur J Nucl Med Mol Imaging. 2024 Sep;51(11):3161-3175. doi: 10.1007/s00259-024-06743-5. Epub 2024 May 7. PMID 38713298
- [Background] Zhang Y, Wang Y, Chen Y, Ding X, Wang S, Liu W, Hu M, Liu Z. PET Imaging of Peptide Probe Al[18F]F-NOTA-PCP1 for Monitoring the Engagement of PD-L1 Antibodies in Tumors. Mol Pharm. 2024 Mar 4;21(3):1515-1525. doi: 10.1021/acs.molpharmaceut.3c01151. Epub 2024 Jan 30. PMID 38291578